CLINICAL TRIAL: NCT06302920
Title: Investigation of the Effect of Kinesiotaping on Pain, Swelling and Kinesiophobia in Patients Diagnosed With Complex Regional Pain Syndrome
Brief Title: Effect of Kinesiotaping on Pain,Edema and Kinesiophobia in Patients With Complex Regional Pain Syndrome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alanya Alaaddin Keykubat University (Other)
Responsible Party: Principal Investigator, Deniz Bulut, assistant professor, Alanya Alaaddin Keykubat University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0001
Record Dates: First submitted 2024-02-07; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Complex Regional Pain Syndrome Type I
Keywords: complex regional pain syndrome; kinesiotaping; Kinesiophobia
MeSH Terms: conditions — Complex Regional Pain Syndromes; Kinesiophobia | interventions — Athletic Tape

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Kinesiotaping group (Active Comparator): Patients will be divided into 2 groups according to the random numbers table, and both groups will receive a conventional physical therapy and rehabilitation program and nutritional support. Afterwards, edema-reducing kinesiotaping will be applied to one group.
  Interventions: Device: Kinesiotape
- Control group (No Intervention): Patients will be divided into 2 groups according to the random numbers table, and both groups will receive a conventional physical therapy and rehabilitation program and nutritional support.

INTERVENTIONS:
Device: Kinesiotape — Lymphatic correction technique
  Arms: Kinesiotaping group

SUMMARY:
Patients will be divided into 2 groups according to the random numbers table, and both groups will receive a conventional physical therapy and rehabilitation program and nutritional support. Afterwards, edema-reducing kinesiotaping will be applied to one group. The applied kinesio tape will remain on the patient for 5 days and will be taped again after 2 days without tape. In this way, taping will be done 3 times in total, once a week for 3 weeks. During this period, patients will continue their routine physical therapy program and measurements will be taken by the same researcher in the 1st week of treatment and 3 weeks later.

DETAILED DESCRIPTION:
Patients will be divided into 2 groups according to the random numbers table, and both groups will receive a conventional physical therapy and rehabilitation program and nutritional support. Afterwards, edema-reducing kinesiotaping will be applied to one group. The applied kinesio tape will remain on the patient for 5 days and will be taped again after 2 days without tape. In this way, taping will be done 3 times in total, once a week for 3 weeks. During this period, patients will continue their routine physical therapy program and measurements will be taken by the same researcher in the 1st week of treatment and 3 weeks later.

Kinesiology tapes have a wavy structure in line with the structure and physiological functions of the skin and have adhesive properties. The adhesive is a heat-activated acrylic. After approximately 20 minutes, the adhesive is fully activated. The tapes are porous, permeable to air and liquid, allow perspiration and dry quickly.Kinesiology tapes have a wavy structure in line with the structure and physiological functions of the skin and have adhesive properties. The adhesive is a heat-activated acrylic. After approximately 20 minutes, the adhesive is fully activated. The tapes are porous, permeable to air and liquid, allow perspiration and dry quickly. The method of application varies depending on the cutting method, application direction and region of the tape. If the anatomy of muscles, joints, ligaments and circulatory system is mastered and the correct techniques appropriate to the situation are used, the chance of success of the technique increases. Lymphatic correction technique is used to reorganize damaged lymphatic circulation. The main goals are to create a dead space in the tissue that allows circulation and to reduce the pressure on the lymph vessels at the tissue level. It directs lymph fluid to larger lymphatic vessels and lymph nodes. This effect can be explained by the elastic qualities and lifting effect of the tape. While lifting the surface skin reduces pressure and ensures lymphatic circulation, the tape provides a massage effect during active movement. Thanks to the tape, maximum contraction and relaxation of the muscles is ensured and the effectiveness of the deeper lymphatic flow is increased.

Kinesiophobia (also known as fear of movement); It is defined as an excessive and irrational fear of physical movement to avoid being harmed or injured again. It can also be expressed as an excessive, irrational fear of physical movement and activity resulting from a feeling of vulnerability due to pain. Its prevalence in chronic pain varies between 50-70%. While the existing threatening characteristics of the pain experience may vary depending on the situation and the person, avoidance behavior, which is protective in the short term, paradoxically worsens the problem in the long term. It is stated that kinesiophobia is an important factor in the transition of pain from acute to chronic stages.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of reflex sympathetic dystrophy Ability to be included in a physical therapy program

Exclusion Criteria:

Hemiplegia Malignancy Polyacrylamide allergy Open wound in the area to be applied

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-05-20 (Estimated); Primary Completion 2024-06-20 (Estimated); Study Completion 2024-12-20 (Estimated)

PRIMARY OUTCOMES:
Resting pain | Beginning, week 3 and week 6
  The resting pain level of the patients will be measured with the Visual Analogue Scale (VAS).A score between 0 and 10 will be determined by the patient, with 0 being no pain and 10 being the most severe pain level.
Edema | Beginning, week 3 and week 6
  The patients will be physically examined and their wrist circumference and metacarpal circumference will be measured in centimeters.
Kinesiophobia | Beginning, week 3 and week 6
  Kinesiophobia will be assessed using the Tampa Scale for Kinesiophobia. A score above 37 in the test is defined as an indicator of a high level of kinesiophobia.

CONTACTS AND LOCATIONS:
Overall Officials: Deniz Bulut, A.professor, Principal Investigator — Alanya Alaaddin Keykubat University
Locations (1):
- Alanya Alaaddin Keykubat University, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fischer SGL, Zuurmond WWA, Birklein F, Loer SA, Perez RSGM. Anti-inflammatory treatment of Complex Regional Pain Syndrome. Pain. 2010 Nov;151(2):251-256. doi: 10.1016/j.pain.2010.07.020. Epub 2010 Aug 7. No abstract available. PMID 20692766
- [Background] Çeliker R, Güven Z, Aydoǧ T, et al. Kinezyolojik bantlama tekniǧi ve uygulama alanlari. Turkiye Fiz Tip ve Rehabil Derg. 2011;57(4):225-235.
- [Background] Roelofs J, van Breukelen G, Sluiter J, Frings-Dresen MHW, Goossens M, Thibault P, Boersma K, Vlaeyen JWS. Norming of the Tampa Scale for Kinesiophobia across pain diagnoses and various countries. Pain. 2011 May;152(5):1090-1095. doi: 10.1016/j.pain.2011.01.028. PMID 21444153